CLINICAL TRIAL: NCT03588052
Title: Evaluation of Esthetic Root Coverage Using Platelet-Rich Fibrin Versus Subepithelial Connective Tissue Graft With Vestibular Incision Subperiosteal Tunnel Access Technique in Patients With Multiple Gingival Recessions: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Esthetic Root Coverage Using Platelet-Rich Fibrin Versus Subepithelial Connective Tissue Graft With Vestibular Incision Subperiosteal Tunnel Access in Multiple Gingival Recessions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Medhat Sery, B.Sc. in Oral and Dental Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4061989
Record Dates: First submitted 2018-06-25; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Gingival Recession
Keywords: Vestibular incision subperiosteal tunnel access, Subepithelial connective tissue graft, Platelets rich fibrin, Multiple gingival recessions
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VISTA using PRF (Experimental): Vestibular incision subperiosteal tunnel access combined with Platelets-Rich Fibrin
  An intravenous blood will be drawn from the patient in a glass-coated plastic tubes, centrifuged at 3000 rpm for 10-12 min. A Platelets rich fibrin membrane will then be obtained
  Interventions: Procedure: VISTA using PRF
- VISTA using SCTG (Active Comparator): vestibular incision subperiosteal tunnel access combined with subepithelial connective tissue graft
  Subepithelial connective tissue graft will be harvested from the palate, secured in the tunnel to cover the root dehiscence then sutured
  Interventions: Procedure: VISTA using SCTG

INTERVENTIONS:
Procedure: VISTA using PRF — Vertical vestibular access incision will be done through the periosteum to elevate a subperiosteal tunnel, exposing the facial osseous plate. The tunnel will be extended beyond mucogingival junction and at least one or two teeth beyond the teeth indicated for root coverage to mobilize gingival margins and allow for low-tension coronal repositioning of the gingiva.
  Freshly prepared platelet-rich fibrin will be secured in the tunnel to cover the root dehiscence, coronal advancement of gingival margin and suturing to the facial aspect of each tooth to avoid apical relapse of the gingival margin during the initial phase of healing. The vertical incision will be then approximated and sutured
  Other Names: Vestibular incision subperiosteal tunnel access technique with Platelet-rich fibrin
  Arms: VISTA using PRF
Procedure: VISTA using SCTG — Vertical vestibular access incision will be done through the periosteum to elevate a subperiosteal tunnel, exposing the facial osseous plate. The tunnel will be extended beyond mucogingival junction and at least one or two teeth beyond the teeth indicated for root coverage to mobilize gingival margins and allow for low-tension coronal repositioning of the gingiva.
  Subepithelial connective tissue graft will be secured in the tunnel to cover the root dehiscence, coronal advancement of gingival margin and suturing to the facial aspect of each tooth to avoid apical relapse of the gingival margin during the initial phase of healing. The vertical incision will be then approximated and sutured
  Other Names: Vestibular incision subperiosteal tunnel access technique with Subepithelial connective tissue graft
  Arms: VISTA using SCTG

SUMMARY:
Patients with gingival recession, complain of excessive tooth length that affects their appearance during smiling or functioning. The main goal of plastic periodontal surgeries is to restore patient's esthetic demands with the regeneration of gingival and periodontal tissues.

Although SCTG is considered a gold standard, it has its own limitations like patient morbidity and graft availability. Consequently, PRF has been introduced in an attempt to overcome the drawbacks of SCTG and achieve optimum results in root coverage.

The minimally invasive VISTA technique allows better access with coronal positioning and stabilization of gingival margin to achieve complete root coverage. In addition to platelets-rich fibrin that gives a predictable and reproducible result in restoring the amount of keratinized tissue, root coverage and better esthetic outcome. The use Vestibular incision subperiosteal tunneling access (VISTA) with platelet-rich fibrin will be used to achieve complete root coverage.

DETAILED DESCRIPTION:
Gingival recession is defined as apical displacement of gingival margin beyond the cementoenamel junction leading to the exposure of root surface. There are various etiologic factors for gingival recession like trauma, infection and other anatomical factors.

Nowadays, periodontal plastic surgeries for treatment of gingival recession have become an important array due to increase in patient's esthetic demands and other conditions such as dentin hypersensitivity, root caries or abrasion, keratinized tissue augmentation and gingival margin discrepancy.

Subepithelial connective tissue grafts (SCTG) are considered the gold standard to obtain maximum root coverage due to its characteristics of quick keratinization and periodontal connective tissue adherence, in addition to its good blood supply to the graft and high degree of gingival color match and esthetics. However, the application of this technique is limited by the thickness of the donor tissue, anatomical factors, limited quantity compromising their use in multiple recession, tissue morbidity, and technique sensitive with postoperative pain, bleeding and swelling.

Accordingly, alternative membranes and new biomaterials have been introduced to overcome the limitations of SCTG.

Platelet rich fibrin (PRF) was introduced; a second generation platelet concentrate. PRF contains growth factors that play an essential role in soft and hard tissue regeneration; they promote fibroblastic proliferation, increase tissue vascularization, enhance soft tissue healing potential and accelerate bone regeneration. These growth factors include (PDGFs), epidermal growth factor (EGF), transforming growth factor beta (TGF-β), vascular endothelial growth factor (VEGF).

Vestibular incision subperiosteal tunnel access (VISTA), a novel minimal invasive technique for achieving root coverage that overcome the limitation of the previous intrasulcular tunneling techniques.

Hence this study will performed to evaluate the use of PRF in conjunction with VISTA technique in management of patients with multiple gingival recessions

ELIGIBILITY:
Inclusion Criteria:

1. Multiple adjacent maxillary or mandibular gingival recessions Miller class І or II
2. Good oral hygiene with full mouth plaque score (FMPS) ≤ 20% (O'Leary et al. 1972)

Exclusion Criteria:

1. Any systemic condition that may contraindicate periodontal surgery
2. Individuals taking medications that interfere with periodontal tissue health or healing
3. Previous periodontal plastic surgery in the selected sites for at least 6 months before the study
4. Pregnancy or lactating women
5. Former or current smokers
6. Active periodontal disease
7. Non-compliant patients.
8. Any restorations found in the selected sites

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-20 (Estimated)

PRIMARY OUTCOMES:
Amount of root coverage | 6 months
  complete root coverage after surgical correction measured in millimeters by using periodontal probe

SECONDARY OUTCOMES:
Root Coverage Esthetic score a numbering score | 6 months
  A scoring system to evaluate esthetics after surgical root coverage giving a numbering score by a periodontal probe
Post-Operative Pain a numerical rating scale | 14 days
  Numerical Rating Scale (NRS) with numbers from 0 to 10 ('no pain' to 'worst pain imaginable')for the first 2 weeks postoperatively.
Post-Operative Swelling verbal rating scale | 7 days
  Verbal Rating Scale (VRS); absent(no swelling), slight (intraoral swelling at the operated area), moderate (moderate intraoral swelling at the operated area) and intense (intensive extraoral swelling extending beyond the operated area)
Post-Surgical Patient Satisfaction numerical rating scale | 14 days
  A numerical rating scale will be used. A 3-item questionnaire is asked and the patients shall use a 7 point answer scale.
Clinical Attachment level gain in millimeters | 6 months
  the clinical attachment level is the measurement of the position of the soft tissue in relation to the cemento-enamel junction (CEJ). Two measurements are used to calculate the CAL: the probing depth and the distance from the gingival margin to the CEJ. measured using a periodontal probe in millimeters.
Probing depth in millimeters | 6 months
  It is measuring the distance from the gingival margin to the base of the pocket using periodontal probe. The probe will be inserted parallel to the long axis of the tooth using light force.
Keratinized Tissue Width in millimeters | 6 months
  It is measured from the free gingival margin to the mucogingival junction (MGJ). By using the periodontal probe, MGJ will be identified using the roll technique
Gingival Thickness in millimeters | 6 months
  It is measured by penetrating the gingiva mid-buccally in the attached gingiva, half way between mucogingival junction and free gingival groove to measure the gingival thickness

CONTACTS AND LOCATIONS:
Overall Officials: Mona Darhous, Phd, Study Director — Cairo University; Ahmed El-Barbary, Phd, Study Chair — Cairo University; Marwa Hegab, Phd, Study Chair — Cairo University; Yasmin Sery, Bachelor, Principal Investigator — Cairo University